CLINICAL TRIAL: NCT06796582
Title: Agreement of the Estimated 1-Repetition-Maximum Between Two Multiple-Repetition-Maximum Tests with Different Weight in Patients with Cardiovascular Disease or Risk Factors
Brief Title: Reliability of Multiple-Repetition-Maximum Tests in Patients with Cardiovascular Disease or Risk Factors
Status: Not yet recruiting | Type: Observational
Sponsor: Technical University of Munich (Other)
Responsible Party: Principal Investigator, Stephan Mueller, Exercise Physiologist (Postdoctoral Researcher), Technical University of Munich
Other Study IDs: 2025-27-S-CB
Record Dates: First submitted 2025-01-22; First posted 2025-01-28 (Actual); Last update posted 2025-01-29 (Actual); Status verified 2025-01

CONDITIONS: Heart Failure; Coronary Heart Disease (CHD); Atrial Fibrillation (AF); Diabetes Mellitus; Arterial Hypertension
Keywords: resistance training; cardiovascular disease; cardiovascular risk factors; muscle strength
MeSH Terms: conditions — Heart Failure; Coronary Disease; Atrial Fibrillation; Diabetes Mellitus; Hypertension; Cardiovascular Diseases

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
Exercise training is a cornerstone in the prevention and rehabilitation of cardiovascular disease. While research has primarily focused on endurance training, resistance training becomes more and more important. The gold standard to prescribe resistance training intensity or monitor longitudinal changes is the 1-Repetition-Maximum (1-RM) test. However, particularly for unexperienced individuals, this test may not be recommendable due to the high load and an increased risk of injuries. Alternatively, there are several published formulas to estimate the 1-RM based on a multiple-repetition-maximum (or repetition-to-failure) test. However, these formulas have been primarily tested in healthy individuals. Moreover, the reliability of the 1-RM estimation based on two tests with different submaximal weight is unknown. Therefore, the present study evaluates the agreement of the 1-RM estimation (based on different formulas) between two Multiple-RM tests with different weight in 50 patients with cardiovascular disease (heart failure, coronary heart disease, atrial fibrillation) or cardiovascular risk factors (type 2 diabetes, arterial hypertension).

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 50 years
* At least one of the following cardiovascular diseases / risk factors:
* Heart failure
* Coronary heart disease
* Atrial fibrillation
* Arterial hypertension
* Type 2 diabetes mellitus
* Clinically stable for ≥ 4 weeks
* Medical clearance to perform resistance training / strength testing
* Signed written informed consent

Exclusion Criteria:

* Pregnancy
* Acute infection
* Chronic joint inflammation
* Knee, hip, ankle, wrist, elbow or shoulder pain
* Known osteoporosis (T-value ≤ -2.5)
* Uncontrolled hypertension (≥160 mmHG systolic / ≥100 mmHG diastolic)
* Known cerebral or thoracic aneurysm

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who visit the outpatient clinic for Preventive Sports Medicine and Sports Cardiology at the TUM University Hospital, Munich, Germany
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2025-02 (Estimated); Primary Completion 2025-06 (Estimated); Study Completion 2025-06 (Estimated)

PRIMARY OUTCOMES:
Estimated 1-Repetition-Maximum | cross-sectional study (day 1)
  The estimated 1-Repetition-Maximums based on two Multiple-Repetition-Maximum tests with different weight will be compared using Bland-Altman plots. Acceptable Limits of Agreement are defined as +/- 10%. The comparisons will be performed using different published formulas to evaluate, which formula(s) may be recommended in patients with cardiovascular disease / risk factors. The study will be performed on the following resistance training machines: leg press and chest press

SECONDARY OUTCOMES:
Number of repetitions required to perform a valid Multiple-Repetition-Maximum test | cross-sectional (day 1)
  The Multiple-Repetition-Maximum test is considered valid if muscular failure occurs after completion of 2-10 repetitions. This is based on the evidence that (most) published formulas become less precise if >10 repetitions can be performed.
Adverse Events | cross-sectional (day 1)
  any adverse events that occur in relation to the Multiple-Repetition-Maximum Tests will be documented

CONTACTS AND LOCATIONS:
Overall Officials: Stephan Mueller, Dr rer nat, Principal Investigator — Technical University of Munich, Department for Preventive Sports Medicine and Sports Cardiology

IPD SHARING:
Plan to Share IPD: Undecided
Data sharing will depend on the possibility to anonymize the requested data set and must be approved by the data security department of the TUM University Hospital